CLINICAL TRIAL: NCT03749369
Title: Effect of Salvadora Persica on Clinical, Radiographic and Microbiological Parameters of Chronic Periodontitis: A Triple-Blind Randomized Controlled Clinical Trial
Brief Title: Adjunctive Use of Salvadora Persica in Chronic Periodontitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Collaborators: Ziauddin University (Other)
Responsible Party: Principal Investigator, Zohaib Akram, Senior Registrar, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZCD
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP plus salvadora persica root (Active Comparator): Subjects receiving salvadora gel in addition to scaling and root planing
  Interventions: Drug: Salvadora Persica Root; Procedure: Scaling and root planing
- SRP only (Placebo Comparator): Subjects receiving scaling and root planing only
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Drug: Salvadora Persica Root — Salvadora Persica Gel
  Other Names: SP gel
  Arms: SRP plus salvadora persica root
Procedure: Scaling and root planing — Thorough scaling and root planing (SRP) will be performed by a single clinician. The SRP procedure will be carried out in two sittings, comprising of ultrasonic scaling in the first, and manual instrumentation and root debridement in the second.
  Other Names: SRP

SUMMARY:
A randomized controlled triple blinded study to evaluate the effectiveness of Salvadora Persic (SP) as an adjunct to Scaling and Root Planing (SRP) in chronic periodontitis by comparing the basic parameters of periodontitis, radiographs and bacterial levels with a controlled group (SRP only).

DETAILED DESCRIPTION:
Sixty-six subjects with untreated, moderate-to-severe chronic periodontitis will be selected by convenience sampling. The participants will be randomly divided into 2 groups:

1. Test group: SRP + SP gel
2. Control group: SRP only

Each participant will undergo treatment in the following steps:

1. QUESTIONNAIRE:

   All participants will complete a structured baseline questionnaire provided by one trained interviewer that will include the data regarding; (a) age; (2) gender; (3) education status; (4) occupation; (5) medical status
2. INFORMED CONSENT:

   All eligible subjects will be thoroughly informed of the nature, potential risks and benefits of their participation in the study.
3. ASSESSMENT OF PARAMETERS:

   1. CLINICAL PERIODONTAL PARAMETERS Full-mouth plaque index (PI), bleeding on probing (BOP), probing depth (PD), and clinical attachment loss (CAL) will be recorded on baseline, 6th week and 12th week for all the patients that pass the inclusion criteria.
   2. RADIOGRAPHIC ANALYSIS The depth of bony defects (BD) will be evaluated at baseline, 6 and 12 weeks using image analysis software (Scion Image Analyzer, Scion, Frederick, MD, USA).
   3. ANALYSIS OF PLAQUE MICROORGANISM Subgingival plaque will be collected at baseline and 12 weeks from the deepest PD (>4mm) of each patient.
4. SCALING AND ROOT PLANING After baseline recordings, thorough SRP will be performed by a single clinician. The SRP procedure will be carried out in two sittings, comprising of ultrasonic scaling in the first, and manual instrumentation and root debridement in the second.
5. APPLICATION OF SP GEL In the test group, areas with PPD greater than 4 mm will be marked on the periodontal chart. In these areas SP gel will be placed following root planing procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are >30 years old
2. Minimum of 20 teeth , excluding third molars
3. Systemically healthy patients with moderate (PD of 5 to 6 mm or clinical attachment loss CAL of 4 to 6 mm) or deep pockets (PD ≥7mm or CAL of 6 to 9 mm) and vertical bone loss ≥3 mm on intraoral periapical radiographs (Armitage 1999)

Exclusion Criteria:

1. Presence of systemic conditions that could modify the progression of periodontitis such as diabetes mellitus, metabolic syndrome, cardiovascular disease or immunologic disorders
2. Systemic antimicrobials in the previous 6 months
3. Aggressive periodontitis
4. Pregnancy or lactation
5. Inability to provide informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
clinical attachment level | 3 months
  Clinical attachment level (CAL) is the distance from the cemento-enamel junction to the base of the sulcus. It will be measured by a calibrated examiner who will use a UNC 15 probe at 6 points around each tooth. The measurements will be expressed as the nearest millimeters and will be entered into the advanced periodontal chart.
periodontal pocket depth | 3 months
  Probing depth (PD) is defined as the distance from the gingival margin to the base of the pocket/sulcus.It will be measured by a calibrated examiner, using a UNC 15 probe and expressed in millimetres. The value will be entered into the periodontal chart provided with the questionnaire.
bleeding on probing | 3 months
  presence or absence of bleeding on probing within 10 seconds around 6 points along each tooth. Presence of bleeding will be marked as 1, while absence will be marked as 0.
plaque index | 3 months
  presence of absence of plaque along 6 points around each tooth will be examined and entered in the periodontal chart. SItes showing plaque will be marked as 1, while those not showing plaque will be marked as 0.

SECONDARY OUTCOMES:
intrabony defects | 3 months
  Bony defects will be measured on the radiograph by measuring the distance from the cemento-enamel junction to the crest of the bone.
Porphyramonas gingivalis level | 3 months
  assessment of porphyromona ginivalis levels will be done utilising the Real-time Polymerase Chain Reaction (PCR) at baseline and 3 months.

IPD SHARING:
Plan to Share IPD: Undecided